CLINICAL TRIAL: NCT03147365
Title: Aerobic Training Versus Strength Exercises on Quality of Life and Functional Capacity on Children With Leukemia.
Brief Title: Effect of Different Exercises on Quality of Life of Leukemia Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Cancer Hospital Egypt 57357 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CCHE-ALL003
Record Dates: First submitted 2017-04-02; First posted 2017-05-10 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-01

CONDITIONS: Quality of Life; Acute Lymphoblastic Leukemia; Exercise
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Experimental controlled randomization using Block Stratified Randomized Software program, after obtaining informed consent from illegible patient or his caregiver.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Twenty five children who will not receive any physical therapy treatment.
- Study group A (Experimental): Twenty five children who will receive physical therapy treatment which include aerobic exercises.
  Interventions: Behavioral: Aerobic exercises
- Study group B (Experimental): Twenty five children who will receive physical therapy treatment which include modified strength training program.
  Interventions: Behavioral: Modified strength training

INTERVENTIONS:
Behavioral: Aerobic exercises — Aerobic exercises will do by using treadmill for children of study group A. it will consist of (max.incline15% - max. speed - heart rate grips and wireless chest strap - smooth virtual fitness trainer - smooth drop folding frame - impression shock absorption cushioning system).
  Arms: Study group A
Behavioral: Modified strength training — Dumbbells will be used to conduct the modified strength training program for children of group B. This exercises included five exercises for the main muscle groups: bench press, leg press, seat row, leg extension and lat pull down.
  Arms: Study group B

SUMMARY:
* To compare between modified strength training program and aerobic exercises on quality of life on children with Acute Lymphoblastic Leukemia.
* To compare between modified strength training program and aerobic exercises on functional capacity on children with Acute Lymphoblastic Leukemia.

DETAILED DESCRIPTION:
This study will be done to determine any exercise from aerobic exercises or modified strength training program will be more effective on quality of life and functional capacity on children with Acute Lymphoblastic Leukemia .Acute Lymphoblastic Leukemia is wide spread in the world and the children with this disease are fragile so must know the most program effect.

ELIGIBILITY:
Inclusion Criteria:

* Age range from8-12years.
* Children during 3rd phase( maintenance phase of the treatment). According San et al(2007) who found children with Acute Lymphoblastic Leukemia in maintenance phase of treatment can safely perform both aerobic and resistance training .
* Time elapsed since the start of the maintenance phase >20weeks.
* Children with muscle weakness due to chemotherapy.
* The height , weight and body mass index of the child will take on standard scale.
* preserved cardiac structure and function as assisted by echo-cardiogram.
* The children have ability to walk.

Exclusion Criteria:

Children who have one or more of the following criteria will be excluded from the study:

* Receiving more intensive chemotherapy.
* Mental disabled.
* Sever cardiomyopathy (ejection fraction <40%, ECG will be used as a pretest as it might be a more sensitive tool to exclude angina pectoris).
* Low blood platelet levels (< 50.000 per µl).
* Marked anemia (hemoglobin < 8 g/dl).
* Severe cachexia (i.e., weight mass loss > 35%).
* Pain in bone.
* Inability to walk.
* Sensory disturbance.
* Peripheral neuropathy.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2017-03-05 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2020-04-05 (Actual)

PRIMARY OUTCOMES:
Improvement of quality of life | at week 20
  The pediatric quality of life inventory (PedsQL) is a modular approach to measure health-related quality of life in healthy children and adolescents and those with acute and chronic health conditions.

SECONDARY OUTCOMES:
Improvement of functional capacity | at week 20
  6 minute walk test is a test to measure functional capacity by using pulse oximeter to detect percentage of oxygen saturation at peripheral capillaries.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa M Khalifa, BSc, Principal Investigator — Children's Cancer Hospital Egypt CCHE 57357
Locations (1):
- Children's Cancer Hospital Egypt 57357, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No